CLINICAL TRIAL: NCT04855877
Title: Does Oral Administration of Tranexamic Acid in Anterior Cruciate Ligament Arthroscopic Surgery Reduce Postoperative Haemarthrosis and Improve Functional Prognosis?
Brief Title: Oral Administration of Tranexamic Acid in Anterior Cruciate Ligament Surgery Reduce Postoperative Haemarthrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of Anesthesiology Departement, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TRANEX-LCA
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Hemorrhage Postoperative; Anterior Cruciate Ligament Rupture; Arthroscopy; Total Blood Loss
MeSH Terms: conditions — Postoperative Hemorrhage; Anterior Cruciate Ligament Injuries; Exsanguination | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Double blinded prospective randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, anesthesiologist and surgeon are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Tranexamic Acid (Active Comparator): 52 patients scheduled for primary anteriori cruciate ligament surgery by arthroscopy
  Interventions: Drug: Oral tablet
- Placebo (Placebo Comparator): 52 patients scheduled for primary anteriori cruciate ligament surgery by arthroscopy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral tablet — Oral administration of 2 grammes tranexamic acid 2 hours before skin incision and 2 grammes oral tranexamic acid 4 hours after first administration
  Arms: Oral Tranexamic Acid
Drug: Placebo — Oral administration of lactose tablet (placebo)
  Arms: Placebo

SUMMARY:
To find superiority relationship between oral and intravenous administration of tranexamic acid on peroperative and postoperative blood loss, haemarthrosis prevalence and improvement functional prognosis in anterior cruciate ligament arthroscopy.

DETAILED DESCRIPTION:
Tranexamic acid is an anti-fibrinolytic drug, recommended in total hip arthroplasty to reduce peroperative and postoperative hemorrhagic complications. The original character of our study lies in the serum dosage of tranexamic acid, allowing to correlate the primary objective (blood loss) with this one. The investigators will focus on the reduction of the risks associated with the administration of intravenous medicines, the economic aspect and the ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Primary arthroscopic surgery for anterior cruciate ligament reconstruction

Exclusion Criteria:

* Renal failure with serum creatinine level higher than 1,40 mg/dL
* Thromboembolic events in last 12 months before surgery
* Pregnancy
* Congenital or acquired coagulation diseases
* History of gastric surgery that could lead to malabsorption
* Diabetic gastro-paresis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of haemarthrosis | First 24 hours after surgery
  Postoperative (drainage) blood loss

SECONDARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Postoperative pain score on numeric ratio scale (NRS) from 0 (no pain) to 10 (worst pain)
Postoperative pain | 72 hours after surgery
  Postoperative pain score on numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain)
Postoperative pain | 7 days after surgery
  Postoperative pain score on numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain)
Postoperative pain | 15 days after surgery
  Postoperative pain score on numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain)
Clinical evaluation of functional recovery | 1 days after surgery
  Tegner activity score from 0 (no activity) to 10 (competitive sport)
Clinical evaluation of functional recovery | 3 days after surgery
  Tegner activity score from 0 (no activity) to 10 (competitive sport)
Clinical evaluation of functional recovery | 7 days after surgery
  Tegner activity score from 0 (no activity) to 10 (competitive sport)
Clinical evaluation of functional recovery | 15 days after surgery
  Tegner activity score from 0 (no activity) to 10 (competitive sport)
Length of hospital stay | First 30 days after surgery
  Total days of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. Tranexamic acid in total joint arthroplasty: the endorsed clinical practice guides of the American Association of Hip and Knee Surgeons, American Society of Regional Anesthesia and Pain Medicine, American Academy of Orthopaedic Surgeons, Hip Society, and Knee Society. Reg Anesth Pain Med. 2019 Jan;44(1):7-11. doi: 10.1136/rapm-2018-000024. No abstract available. PMID 30640647
- [Background] Muhunthan K, Balakumar S, Navaratnaraja TS, Premakrishna S, Arulkumaran S. Plasma Concentrations of Tranexamic Acid in Postpartum Women After Oral Administration. Obstet Gynecol. 2020 Apr;135(4):945-948. doi: 10.1097/AOG.0000000000003750. PMID 32168220
- [Background] Karaaslan F, Karaoglu S, Yurdakul E. Reducing Intra-articular Hemarthrosis After Arthroscopic Anterior Cruciate Ligament Reconstruction by the Administration of Intravenous Tranexamic Acid: A Prospective, Randomized Controlled Trial. Am J Sports Med. 2015 Nov;43(11):2720-6. doi: 10.1177/0363546515599629. Epub 2015 Sep 2. PMID 26337246